CLINICAL TRIAL: NCT06200896
Title: Single-Center, Two- Arm Study to Evaluate the Safety and Device Functionality of the SFM Anastomosis Device and Delivery System, When Used to Create a Duodenal-Ileal Anastomosis to Revise a Post SG (SNAP-PS), or Used to Create a Jejuno-Jejunal (J-J) Anastomosis of a Roux-en-Y
Brief Title: Early Feasibility Study: Assessment of Self-Forming Magnetic Anastomosis Device and Delivery System (SFM) in Obese Patients, When Used to Create a Duodenal-Ileal Anastomosis Post SG (SNAP-PS), or Used to Create a Jejuno-Jejunal (J-J) Anastomosis
Acronym: GIW-J-J
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIW 23-004
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SFM in Obese Patients, When Used to Create a Duodenal-Ileal Anastomosis Post Sleeve Gastrectomy (Experimental): Duodenal-Ileal Anastomosis Post Sleeve Gastrectomy created with Self Forming Magnets (SFM)
  Interventions: Device: Self Forming Magnets used to Create A Compression Anastomosis
- SFM in Obese subjects when Used to Create a Jejuno-Jejunostomy (J-J) Anastomosis (Experimental): Jejuno-Jejunostomy (J-J) Anastomosis created with Self Forming Magnets (SFM) as part of a Roux-en-Y gastric bypass
  Interventions: Device: Self Forming Magnets used to Create A Compression Anastomosis

INTERVENTIONS:
Device: Self Forming Magnets used to Create A Compression Anastomosis — Self Forming Magnets used to Create A Compression Anastomosis connecting the Duodenum to the ileal in Post Sleeve Gastrectomy Patients and Jejunum to jejunum in Roux-en-Y patients.

SUMMARY:
The objectives of this study are to assess the initial safety and device functionality of the SFM Anastomosis System including delivery systems when used to create a duodenal-ileal (D-I) anastomosis with patients with prior sleeve gastrectomy who experience inadequate weight loss (i.e., SNAP-PS procedure). Additionally, the study is designed to evaluate the potential of the SFM Anastomosis System to create a Jejuno-jejunostomy in Roux-en-Y gastric bypass procedures.

DETAILED DESCRIPTION:
This is a two-arm, single-center, early feasibility study to evaluate the use of the SFM Anastomosis System for creation of a duodenal-ileal (D-I) anastomosis in participants who have experienced inadequate weight loss following sleeve gastrectomy (SNAP-PS cohort) defined to be failure to achieve a minimum 50% EWL post sleeve gastrectomy or a patient undergoing a Roux-en-Y gastric bypass the SFM will be used to create the jejuno-jejunostomy. Adult male and female subjects between the ages of 18 and 65 years-old who are candidates for the primary or revisional surgery will be considered for participation.

Patients appearing to meet basic eligibility criteria and who sign the study specific consent form will be screened for enrollment into this study and will be assessed by a multidisciplinary research team with pre-procedure nutritional and medical evaluation (including psychological and behavioral evaluation by an internist/bariatrician).

Subjects meeting the inclusion and exclusion criteria and enrolled into the study will undergo a procedure in which the SFM device and delivery systems with create anastomoses between the duodenum and ileum or jejunum to jejunum.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years at screening
2. For the post sleeve gastrectomy diversion procedures (SNAP-PS)- Obesity with Body Mass Index (BMI) ≥ 40 kg/m2 but ≤ 55 kg/m2 at time of screening with or without comorbidities at time of screening. If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled..
3. For the Roux-en-Y gastric bypass jejuno-jejunostomy procedure (J-J) - Obesity with Body Mass Index (BMI) ≥ 35.1 kg/m2 but ≤50 kg/m2 with or without comorbidities at time of screening. If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled.
4. Able to understand and sign informed consent document
5. Patient lives, and intends to remain, within a 150-km radius of study center for 24 months
6. Willing to commit to sustained healthy behaviors that include diet, eating and exercise habits for the duration of the trial
7. Willing to refrain from smoking during the study follow-up period
8. If subject is female, she must commit to not becoming pregnant for 24 months and agree to use of contraceptives during this period and may not be nursing

Exclusion Criteria:

1. Known or suspected allergy to nickel, titanium or Nitinol
2. Type 1 Diabetes
3. Uncontrolled T2DM Fasting glucose ≥ 200 mg/dl (11.1 mmol/L) and/or hemoglobin A1c >10 or use of injectable insulin
4. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy
5. Contraindication to general anesthesia
6. Clinically significant finding during procedural endoscopy such as presence of an unhealed ulcers, bleeding lesions, tumors or ischemic or necrotic tissue at target magnet deployment site
7. Congenital or acquired anomalies of the GI tract, including atresias, stenosis, prior obstruction or malrotation
8. Presence of a duodenal diverticulum (>10mm)
9. Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding laparoscopically removed gallbladder), pancreas or right colon
10. History of chronic gastrointestinal disease (e.g., cirrhosis, inflammatory bowel disease) that in the opinion of the Investigator may preclude safe and complete study participation
11. Uncontrolled severe hypertension (blood pressure >160/100mmHg)
12. Pre-existing severe comorbid cardio-respiratory disease (e.g., congestive heart failure, uncontrolled cardiac arrhythmia, coronary artery disease, chronic obstructive lung disease requiring supplemental oxygen, pulmonary embolism, Myocardial Infarction with prior 6 months)
13. Liver biochemistries (ALT and AST) ≥ 3 times the upper limit of normal
14. Uncorrectable coagulation disorder (platelets < 100,000, PT >2 seconds above upper normal limit or INR >1.5) at time of procedure, Note: management of anti-platelet medications, when applicable, will follow standard practices of the institution
15. Uncorrectable anemia (Hemoglobin < 11 g/dL in women and <12.5 g/dL in men)
16. Specific genetic or hormonal cause of obesity such as Prader -Willi syndrome
17. For females of child-bearing potential: Pregnancy or desire to be pregnant during the study
18. Concurrent condition anticipated to require MR imaging within the first 2 months after the study procedure
19. Diagnosed Bulimia Nervosa or Binge Eating Disorder (using DSM-5 criteria)
20. Physical or mental disability or psychological illness that in the opinion of the Investigator would be a contraindication for bariatric surgery
21. Subject is immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e.,20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents.
22. Subject has an active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound.
23. Subject is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator"
24. Other prior or concurrent conditions that in the opinion of the Investigator would be unlikely to receive clinical benefit from the study procedure or participation in the study may compromise patient safety or study objectives such as the presence/diagnosis of a severe and evolutive life threatening pathology unrelated to obesity including but not limited to: ongoing infection, chronic pancreatitis, severe hepatic dysfunction, or renal dysfunction (GFR <60mL/min/1.73m2)
25. Any form of substance abuse or psychiatric disorder that in the opinion of the investigator could interfere with the conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ability for physician to create a Magnet (SFM) Anastomosis | 2 days
  Ability to create the anastomosis with SFM without the need for open conversion or use of additional laparoscopic/endoscopic anastomoses devices (endoscopic/laparoscopic suture devices or staplers - except for closure of the laparoscopic enterotomy).
Safety of Creating a Magnet (SFM) Anastomosis | 30 days
  "Freedom from anastomosis adverse events" or "FFAAE" within 30 days including American College of Surgeons (ACS) Grade B/C anastomosis leak (requiring active therapeutic intervention/re-laparotomy), anastomotic bleeding, and small bowel obstruction. All adverse events will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Contreras, MD, Principal Investigator — Head of Surgery
Locations (1):
- Clínica Colonial Hospital, Santiago, Santiago Province, Chile

IPD SHARING:
Plan to Share IPD: No